CLINICAL TRIAL: NCT00430495
Title: A Randomized, Double-blind, Placebo-controlled, Multicentre, Phase II Dose-finding Study of Atacicept Given Subcutaneously in Subjects With Rheumatoid Arthritis and Inadequate Response to TNFa Antagonist Therapy
Brief Title: A Phase 2 Dose-finding Study of Atacicept in Subjects With Rheumatoid Arthritis (AUGUST I)
Acronym: AUGUST I
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: EMD Serono (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 27298
Record Dates: First submitted 2007-01-30; First posted 2007-02-02 (Estimated); Results first posted 2016-02-17 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-01

CONDITIONS: Rheumatoid Arthritis
Keywords: atacicept; arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis | interventions — TACI receptor-IgG Fc fragment fusion protein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Atacicept 25 mg (Experimental)
  Interventions: Drug: Atacicept
- Atacicept 75 mg (Experimental)
  Interventions: Drug: Atacicept
- Atacicept 150 mg (Experimental)
  Interventions: Drug: Atacicept
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo matched to atacicept

INTERVENTIONS:
Drug: Atacicept — Atacicept was administered subcutaneously at a dose of 25 milligram (mg) twice a week for initial 4 weeks as loading dose, followed by 25 mg once a week for subsequent 21 weeks.
  Arms: Atacicept 25 mg
Drug: Atacicept — Atacicept was administered subcutaneously at a dose of 75 mg twice a week for initial 4 weeks as loading dose, followed by 75 mg once a week for subsequent 21 weeks.
  Arms: Atacicept 75 mg
Drug: Atacicept — Atacicept was administered subcutaneously at a dose of 150 mg twice a week for initial 4 weeks as loading dose, followed by 150 mg once a week for subsequent 21 weeks.
  Arms: Atacicept 150 mg
Drug: Placebo matched to atacicept — Placebo matched to atacicept was administered subcutaneously twice a week for initial 4 weeks, followed by once a week for subsequent 21 weeks.
  Arms: Placebo

SUMMARY:
This was a double-blind, placebo-controlled, parallel-arm, multicentre, prospective dose-finding trial of the safety and efficacy of atacicept in subjects with active rheumatoid arthritis who had failed a three month therapeutic trial with a tumor necrosis factor alpha (TNFa) antagonist due to lack of efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Rheumatoid arthritis (RA) satisfying American College of Rheumatology (ACR) diagnostic criteria with a disease history of at least one year
2. Male or female greater than or equal to (>=)18-years of age at time of informed consent
3. Active RA as defined by:

   * >=8 swollen joints (66-joint count),
   * >=8 tender joints (68-joint count), and
   * C-reactive protein (CRP) >=10 milligram per liter (mg/L) (central laboratory) and/or erythrocyte sedimentation rate (ESR) >= to 28 millimeter per hour (mm/h)
4. Failure of at least one TNFa antagonist therapy (previously or at the time of screening) as specified in the protocol
5. Other protocol defined inclusion criteria could apply

Exclusion Criteria:

1. Any condition, including laboratory findings or findings in the medical history or pre-trial assessments, that in the opinion of the Investigator constitutes a risk or a contraindication for the subject's participation in the trial or that could interfere with the trial objectives, conduct or evaluation
2. Treatment with biologics aiming at B cell modulation such as rituximab or belimumab within 2 years before study Day 1
3. Any previous treatment with anakinra (Kineret), abatacept (Orencia) or tocilizumab within 3 months before study Day 1
4. Use of etanercept (Enbrel) within 28 days before study Day 1, or of infliximab (Remicade) or adalimumab (Humira) within 60 days before study Day 1
5. Participation in any interventional clinical trial with an unapproved investigational therapy within the 3 months before the start of this study (or within 5 half-lives of the investigated compound before study Day 1, whichever is longer)
6. Other protocol defined exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2006-12; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — EMD Serono, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (2):
- EMD Serono, Rockland, Massachusetts, United States
- Merck/Serono, Canada, Canada

REFERENCES:
- [Derived] Genovese MC, Kinnman N, de La Bourdonnaye G, Pena Rossi C, Tak PP. Atacicept in patients with rheumatoid arthritis and an inadequate response to tumor necrosis factor antagonist therapy: results of a phase II, randomized, placebo-controlled, dose-finding trial. Arthritis Rheum. 2011 Jul;63(7):1793-803. doi: 10.1002/art.30373. PMID 21452293

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 456 subjects were screened, of whom 256 were enrolled and randomized of which 254 received the trial medication and included in Intention to Treat (ITT) population.
Groups:
- Placebo: Placebo matched to atacicept was administered subcutaneously twice a week for initial 4 weeks, followed by once a week for subsequent 21 weeks.
- Atacicept 25 mg: Atacicept was administered subcutaneously at a dose of 25 milligram (mg) twice a week for initial 4 weeks as loading dose, followed by 25 mg once a week for subsequent 21 weeks.
- Atacicept 75 mg: Atacicept was administered subcutaneously at a dose of 75 mg twice a week for initial 4 weeks as loading dose, followed by 75 mg once a week for subsequent 21 weeks.
- Atacicept 150 mg: Atacicept was administered subcutaneously at a dose of 150 mg twice a week for initial 4 weeks as loading dose, followed by 150 mg once a week for subsequent 21 weeks.
Period: Overall Study
Arm/Group | Placebo | Atacicept 25 mg | Atacicept 75 mg | Atacicept 150 mg
Started | 64 | 66 | 62 | 64
Treated | 62 | 66 | 62 | 64
Completed | 50 | 59 | 49 | 60
Not Completed | 14 | 7 | 13 | 4
Not completed — Adverse Event | 2 | 3 | 2 | 0
Not completed — Death | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 4 | 0
Not completed — Protocol Violation | 1 | 0 | 1 | 0
Not completed — Disease Progression | 1 | 1 | 0 | 0
Not completed — Other | 8 | 2 | 5 | 4
Not completed — Randomized but not Treated | 2 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intention-to-treat (ITT) population included all randomized participants who received at least one treatment dose.
Groups:
- Atacicept 25 mg: Atacicept was administered subcutaneously at a dose of 25 mg twice a week for initial 4 weeks as loading dose, followed by 25 mg once a week for subsequent 21 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | Atacicept 25 mg | Atacicept 75 mg | Atacicept 150 mg | Total
Number analyzed (Participants) | 62 | 66 | 62 | 64 | 254
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.1 (12.5) | 53.4 (13.1) | 55.3 (12.0) | 53.5 (10.1) | 53.8 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 54 | 53 | 53 | 211
  Male | 11 | 12 | 9 | 11 | 43

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving American College of Rheumatology 20 Response Based on C-reactive Protein (ACR20-CRP) at Week 26
Description: ACR20-CRP response is defined as greater than or equal to (>=) 20 percent (%) improvement in both tender joint counts (based on a total of 68 joints) and swollen joint counts (based on a total of 66 joints) together with >=20% improvement in at least 3 of the following 5 measures: 1) participant's assessment of pain; 2) participant's global assessment of disease activity; 3) physician's global assessment of disease activity; 4) participant's assessment of physical function; and 5) acute-phase marker (CRP).
Time Frame: Week 26
Population: ITT population included all randomized participants who received at least 1 treatment dose.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Atacicept 25 mg | Atacicept 75 mg | Atacicept 150 mg
Number analyzed (Participants) | 62 | 66 | 62 | 64
percentage of participants | 29.0 | 30.3 | 27.4 | 39.1

2. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 50 Response Based on CRP (ACR50-CRP) at Week 26
Description: ACR50-CRP response is defined as >=50% improvement in both tender joint counts (based on a total of 68 joints) and swollen joint counts (based on a total of 66 joints) together with >=50% improvement in at least 3 of the following 5 measures: 1) participant's assessment of pain; 2) participant's global assessment of disease activity; 3) physician's global assessment of disease activity; 4) participant's assessment of physical function; and 5) acute-phase marker (CRP).
Time Frame: Week 26
Population: ITT population included all randomized participants who received at least 1 treatment dose.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Atacicept 25 mg | Atacicept 75 mg | Atacicept 150 mg
Number analyzed (Participants) | 62 | 66 | 62 | 64
percentage of participants | 6.5 | 13.6 | 11.3 | 10.9

3. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 70 Response Based on CRP (ACR70-CRP) at Week 26
Description: ACR70-CRP response is defined as >=70% improvement in both tender joint counts (based on a total of 68 joints) and swollen joint counts (based on a total of 66 joints) together with >=70% improvement in at least 3 of the following 5 measures: 1) participant's assessment of pain; 2) participant's global assessment of disease activity; 3) physician's global assessment of disease activity; 4) participant's assessment of physical function; and 5) acute-phase marker (CRP).
Time Frame: Week 26
Population: ITT population included all randomized participants who received at least 1 treatment dose.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Atacicept 25 mg | Atacicept 75 mg | Atacicept 150 mg
Number analyzed (Participants) | 62 | 66 | 62 | 64
percentage of participants | 0.0 | 6.1 | 4.8 | 0.0

4. Secondary Outcome: Percentage of Participants Achieving Disease Activity Score in 28 Joints (DAS28) Based on CRP (DAS28-CRP) of Less Than or Equal to (<=) 3.2 at Week 26
Description: DAS28-CRP incorporates non-graded joint counts for tenderness and swelling based on a total of 28 joints, CRP as a marker of inflammation, and a general health assessment using a 100-millimeter (mm) visual analog scale (the participant's global assessment of disease activity). DAS28 ranges between 0 and 10 representing current disease activity. A value above 5.1 represents high disease activity, a value below 3.2 represents low disease activity, and a value below 2.6 represents remission.
Time Frame: Week 26
Population: ITT population included all randomized participants who received at least 1 treatment dose.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Atacicept 25 mg | Atacicept 75 mg | Atacicept 150 mg
Number analyzed (Participants) | 62 | 66 | 62 | 64
percentage of participants | 9.7 (0.95) | 10.6 (0.84) | 9.7 (0.88) | 12.5 (0.84)

5. Secondary Outcome: Percentage of Participants Achieving Disease Activity Score in 28 Joints (DAS28) Based on CRP (DAS28-CRP) of <=2.6 at Week 26
Description: DAS28-CRP incorporates non-graded joint counts for tenderness and swelling based on a total of 28 joints, CRP as a marker of inflammation, and a general health assessment using a 100 mm visual analog scale (the participant's global assessment of disease activity). DAS28 ranges between 0 and 10 representing current disease activity. A value above 5.1 represents high disease activity, a value below 3.2 represents low disease activity, and a value below 2.6 represents remission.
Time Frame: Week 26
Population: ITT population included all randomized participants who received at least 1 treatment dose.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Atacicept 25 mg | Atacicept 75 mg | Atacicept 150 mg
Number analyzed (Participants) | 62 | 66 | 62 | 64
percentage of participants | 1.6 | 6.1 | 4.8 | 4.7

6. Secondary Outcome: Percentage of Participants Achieving Improvement in Health Assessment Questionnaire Disability Index (HAQ-DI) of at Least 0.3 From Baseline at Week 26
Description: The HAQ-DI is a participant-reported assessment of ability to perform tasks in 8 categories of daily living activities: dress/groom; arise; eat; walk; reach; grip; hygiene; and common activities over past week. Each item was scored on 4-point scale from 0 to 3: 0 = no difficulty; 1 = some difficulty; 2 = much difficulty; 3 = unable to do. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score range is 0 to 3 where 0 = least difficulty and 3 = extreme difficulty. Percentage of participants achieving improvement in HAQ-DI of at least 0.3 from baseline at Week 26 was reported.
Time Frame: Week 26
Population: ITT population included all randomized participants who received at least 1 treatment dose. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Atacicept 25 mg | Atacicept 75 mg | Atacicept 150 mg
Number analyzed (Participants) | 38 | 41 | 34 | 48
percentage of participants | 47.4 | 48.8 | 55.9 | 37.5

7. Secondary Outcome: Percentage of Participants With Good or Moderate European League Against Rheumatism (EULAR) Response at Week 26
Description: The EULAR response criteria evaluate change in DAS28 scores represented as "good response", "moderate response", or "no response" considering both the current DAS28 score and the observed improvement from baseline. Participants were considered to have "good" or "moderate" EULAR response if at the time of assessment, their DAS28 score was <=5.1 and the improvement from baseline in their DAS28 score was greater than (>) 0.6; or if at the time of assessment, their DAS28 score was >5.1 and improvement from baseline in their DAS28 score was >1.2.
Time Frame: Week 26
Population: ITT population included all randomized participants who received at least 1 treatment dose.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Atacicept 25 mg | Atacicept 75 mg | Atacicept 150 mg
Number analyzed (Participants) | 62 | 66 | 62 | 64
percentage of participants | 41.9 | 31.8 | 35.5 | 53.1

8. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was defined as any new untoward medical occurrences/worsening of pre-existing medical condition without regard to possibility of causal relationship. An SAE was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect.
Time Frame: Baseline up to Week 38
Population: Safety population included all randomized participants who received at least 1 treatment dose and had safety data following their first dose.
Measure: Number; unit: participants
Arm/Group | Placebo | Atacicept 25 mg | Atacicept 75 mg | Atacicept 150 mg
Number analyzed (Participants) | 62 | 66 | 62 | 64
participants
  AEs | 41 | 49 | 42 | 46
  SAEs | 3 | 9 | 8 | 5

ADVERSE EVENTS:
Time Frame: Baseline up to Week 38
Arm/Group | Placebo | Atacicept 25 mg | Atacicept 75 mg | Atacicept 150 mg
Serious Adverse Events (participants affected / at risk) | 3/62 | 9/66 | 8/62 | 5/64
Other Adverse Events (participants affected / at risk) | 15/62 | 25/66 | 16/62 | 26/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=62) | Atacicept 25 mg (N=66) | Atacicept 75 mg (N=62) | Atacicept 150 mg (N=64)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 1 | 0
Right ventricular failure (Cardiac disorders) | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1
Pyopneumothorax (Infections and infestations) | 0 | 0 | 0 | 1
Relapsing fever (Infections and infestations) | 0 | 1 | 0 | 0
Stenotrophomonas infection (Infections and infestations) | 0 | 0 | 0 | 1
Diverticular perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Basedow's disease (Endocrine disorders) | 1 | 0 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0 | 0
Vasculitis cerebral (Nervous system disorders) | 0 | 0 | 1 | 0
Fibrin D dimer increased (Investigations) | 0 | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1
Fallopian tube cyst (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Prostatic operation (Surgical and medical procedures) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=62) | Atacicept 25 mg (N=66) | Atacicept 75 mg (N=62) | Atacicept 150 mg (N=64)
Upper respiratory tract infection (Infections and infestations) | 4 | 3 | 0 | 8
Urinary tract infection (Infections and infestations) | 3 | 4 | 3 | 5
Nasopharyngitis (Infections and infestations) | 1 | 3 | 1 | 4
Diarrhoea (Gastrointestinal disorders) | 1 | 4 | 6 | 5
Nausea (Gastrointestinal disorders) | 1 | 5 | 4 | 1
Constipation (Gastrointestinal disorders) | 1 | 4 | 1 | 2
Headache (Nervous system disorders) | 4 | 12 | 5 | 3
Hypertension (Vascular disorders) | 5 | 3 | 3 | 2
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to publishing results, Institution and Principal Investigator (PI) must first provide Sponsor with a copy of proposed publication for review at least 30 days prior to submission. If Institution and PI do not agree to modification, they shall so notify Sponsor and postpone submission for additional 60 days to allow Sponsor to seek legal remedies or file patent applications. There is a need for coordinated approach to any publication of results from sites for any multi-site study.